CLINICAL TRIAL: NCT07383233
Title: Clinical Study on the Efficacy and Safety of CD19/BAFF-R in Vivo CAR-T Cell Therapy Targeting Relapsed/Refractory B Cell Acute Leukemia/Malignant Lymphoma
Brief Title: CD19/BAFF-R in Vivo CAR-T Cell Therapy Targeting Relapsed/Refractory B Cell Acute Leukemia/Malignant Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qi deng (Other)
Responsible Party: Sponsor-Investigator, Qi deng, Chief Physician, Tianjin First Central Hospital
Organization: Tianjin First Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XBAP2025-10
Record Dates: First submitted 2026-01-18; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; CAR T Cell Therapy; Acute Leukemia
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/BAFF-R in vivo CAR-T cell therapy (Experimental)
  Interventions: Biological: CD19/BAFF-R in vivo CAR-T cell intravenous infusion

INTERVENTIONS:
Biological: CD19/BAFF-R in vivo CAR-T cell intravenous infusion — CD19/BAFF-R in vivo CAR-T cell intravenous infusion

SUMMARY:
The currently CAR-T cell therapy in clinical practice largely depends on the expansion of CAR-T cells in vivo. However, the in vitro preparation process of CAR-T cells is complex and costly. In vivo CAR-T cell therapy eliminates the need for ex vivo preparation, significantly reducing treatment costs and procedural complexity. It enables immediate use, thereby improving patient accessibility. CD19 is stably overexpressed in more than 90% of B-cell malignancies. BAFF plays a core regulatory role in the survival, maturation, and homeostasis maintenance of B cells. BAFF-R is selectively expressed on the surface of mature B cell subsets and most B-cell malignancies. Currently, BAFF-R-based CAR-T therapy is in preclinical and early clinical research stages, demonstrating promising therapeutic potential, particularly offering a novel treatment option for patients with CD19-negative or drug-resistant B-cell tumors. The use of CD19/BAFF-R in vivo CAR-T cells as a new anti-tumor therapy may provide a new research direction for the treatment of relapsed/refractory B-cell acute leukemia/malignant lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria：

* The diagnosis was confirmed as B-cell acute leukemia/malignant lymphoma. Requirements for prior treatment: Patients with B-cell acute leukemia/malignant lymphoma who failed to achieve PR after first-line therapy or experienced relapse within 12 months after first-line therapy; or those with relapsed/refractory disease after second-line therapy (a standardized chemotherapy regimen plus salvage chemotherapy). During screening, the patient was in a state of disease recurrence or refractory condition: Acute B-cell leukemia: a) Relapse definition: The presence of blast cells (proportion>5%) in peripheral blood or bone marrow after achieving complete remission with a standardized treatment regimen (including hematopoietic stem cell transplantation), or the development of extramedullary disease; b) Refractory definition: Failure to achieve complete remission after at least two courses of standardized induction therapy. B-cell lymphoma: a) Definition of relapse: PD after achieving remission (including partial response (PR) or complete response (CR)) following adequate treatment; b) Definition of refractory: i. No response to the last treatment: PD during/after the last treatment or SD with a duration of less than 6 months; ii. Relapse or progression after ASCT, including: relapse or PD within 12 months after ASCT, and no response to the last treatment (SD or PD) if salvage therapy is administered.
* The subject's predicted survival time is not less than three months.
* Tumor cells confirmed to be CD19/BAFFR positive by Flow Cytometry (FCM) or Immunohistochemistry.
* Patients with relapsed/refractory B-cell acute lymphoblastic leukemia (B-ALL) and relapsed/refractory B-cell lymphoma (B-LY) who have at least one evaluable lesion.
* Age 14-75 years (inclusive), both genders eligible.
* ECOG performance status ≤ 3.
* HGB≥70g/L(transfusion permitted).
* The functions of vital organs need to meet the following conditions: ①Creatinine ≤ 2.5 × ULN or Cockcroft-Gault creatinine clearance > 50 ml/min (excluding decreased serum creatinine clearance due to lymphoma mass compression), Combination with hemodialysis treatment is permitted. ②LVEF≥50%,② Oxygen saturation ≥90%,③ SCr≤2.5ULN,④ALT and AST≤3ULN,TBil≤2ULN. In the investigator's judgment, if organ dysfunction is associated with the current disease, the enrollment decision will be made by the investigator.
* Subjects intending to conceive must agree to use contraception prior to study enrollment and for six months post-study. In the event of pregnancy or suspected pregnancy, they should promptly notify the investigator.
* The subject or guardian understands and signs the Informed Consent Form (ICF).

Exclusion Criteria:

Any of the following conditions will not be eligible for enrolment:

* Severe heart failure with left ventricular ejection fraction (LVEF) < 50%.
* History of severe pulmonary function impairment.
* Concurrent other progressive malignant tumors.
* Concurrent severe infection that cannot be effectively controlled.
* Concurrent severe autoimmune disease or congenital immunodeficiency.
* Active hepatitis (hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) positive with HBV DNA copy number greater than the upper limit of normal at the study center; Anti-HCV positive with HCV-RNA copy number greater than the upper limit of normal at the study center).
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), or syphilis infection.
* History of severe allergy to biological products (including antibiotics).
* Received inactivated vaccines such as influenza vaccine, COVID-19 vaccine within 4 weeks prior to screening, or received live attenuated vaccines (such as measles, varicella vaccines) within 8 weeks.
* Patients with other severe physical or mental illnesses or laboratory abnormalities that may increase the risk of study participation or interfere with study results, and patients considered unsuitable for this study by the investigator.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of CD19/BAFF-R in vivo CAR-T cell therapy in relapsed/refractory B Cell Acute Leukemia/Malignant Lymphoma | up to one month after the CAR-T infusion
  the incidence and severity of immune therapy related toxic reactions (irAEs)
Evaluate the effcacy of CD19/BAFF-R in vivo CAR-T cell therapy in relapsed/refractory B Cell Acute Leukemia/Malignant Lymphoma | one month and three month after the CAR-T infusion
  CR rate on M1 and M3

SECONDARY OUTCOMES:
Cell pharmacokinetics Dynamic indicators | Day7, Day10, Day14, Day28 after the CAR-T infusion
  CAR-T/T% by flow cytometry
long-term efficacy | up to one year after the CAR-T infusion
  OS